CLINICAL TRIAL: NCT03244826
Title: Shared Care: Patient-Centered Management After Hematopoietic Cell Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Gregory A. Abel, MD, Gregory A. Abel. MD, MPH, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 17-253
Record Dates: First submitted 2017-08-03; First posted 2017-08-10 (Actual); Results first posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-03

CONDITIONS: Other Cancer
Keywords: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Shared Care (Experimental): * For the first 90 days, patients alternate between local oncologist and DFCI for weekly visits.
  * From 90 to 180 days, patients alternate between local and DFCI every 2-3 weeks.
  * Shared Care include the following
    * Formal Care Coordination Plan
    * Patient Engagement and Education
    * Local Oncologist Engagement and Education
    * Patient/Local Oncologist/Transplant Oncologist Web Portal
  Interventions: Other: Shared Care
- Usual Care (Other): * Patients receive all follow-up care at DFCI only, which is currently the Standard Care.
  * Majority of routine visits in first 180 days will be at DFCI.
  Interventions: Other: Standard Care
- Non-Randomized (Other): Patients receive all follow-up care at DFCI only (Standard Care).
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Shared Care — Shared Care involves four specific strategies to allow patients to have a portion of their care locally after HCT, where clinic and laboratory visits are equally shared between the local oncologist and primary HCT team
  Arms: Shared Care
Other: Standard Care — The usual care provided by the transplant center at DFCI.
  Arms: Non-Randomized; Usual Care

SUMMARY:
This research study aims to evaluate the effectiveness of allowing patients who have had a hematopoietic cell transplant to receive some of their post-transplant care with a local oncologist rather than returning to the transplant center for all of their follow-up.

DETAILED DESCRIPTION:
Hematopoietic Cell Transplantation (HCT) - also known as bone marrow transplant - is only available at select centers in the United States which can collect and store stem cells, as well as care for patients before their new immune system cells take hold. For this reason, many patients who undergo HCT live at great distances from their HCT center. Also, after hospital discharge, the first 180 days post-HCT are very important, as patients must be managed closely with frequent follow-up visits.

A potential way to make life easier for HCT patients is to allow some of the post-transplant care to be provided by local oncologists who practice closer to where patients live. This could reduce the burden on patients and their caregivers; however, it is not known if a shared care model would ultimately benefit them. The investigators want to assess the effectiveness of a Shared Care program which allows patients to receive half of their post-HCT care at the HCT center, and the other half with their local oncologist

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years of age
* Scheduled to receive an allogeneic HCT at the Dana-Farber Inpatient Hospital or BWH under the care of a DFCI physician
* Residence in New York, Maine, New Hampshire, Vermont, Connecticut, or Massachusetts
* Referred from or live less than 1 hour from one of the local participating centers.
* Ability to read English (to fill out standard QOL forms)

Exclusion Criteria:

* Age <18 years of age
* Scheduled to receive an autologous HCT
* Has received an allogeneic transplant in the past; scheduled to receive a second allogeneic transplant
* Did not receive an allogeneic HCT at Dana-Farber
* Does not live in New York, Maine, New Hampshire, Vermont, Connecticut, or Massachusetts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A. Abel, MD MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (9):
- United States (9):
  - Stamford Hospital, Stamford, Connecticut
  - Northern Light Cancer Center dba Eastern Maine Medical Center, Bangor, Maine
  - New England Cancer Specialists, Brunswick, Maine
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber at Milford, Milford, Massachusetts
  - Dana-Farber at South Shore Hospital, Weymouth, Massachusetts
  - Dana-Farber at Londonderry, Londonderry, New Hampshire
  - New York Oncology Hematology, Albany, New York
  - Lifespan Cancer Institute at Rhode Island Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abel GA, Kim HT, Zackon I, Alyea ET, Bailey AS, Winters JP, Meehan KR, Reagan JL, Walsh JH, Walsh TP, Ivanov A, Faggen MA, Sinclair S, Joyce AC, Close SD, Emmert A, Koreth J, Antin JH, Cutler CS, Ho VT, Soiffer RJ. Shared Local Oncology Care After Allogeneic Hematopoietic Cell Transplantation: A Randomized Clinical Trial. JAMA Oncol. 2025 Mar 1;11(3):268-275. doi: 10.1001/jamaoncol.2024.5786. PMID 39786764

RESULTS

PARTICIPANT FLOW:
Groups:
- Shared Care: * For the first 90 days, patients alternate between local oncologist and DFCI for weekly visits.
  * From 90 to 180 days, patients alternate between local and DFCI every 2-3 weeks.
  * Shared Care include the following
    * Formal Care Coordination Plan
    * Patient Engagement and Education
    * Local Oncologist Engagement and Education
    * Patient/Local Oncologist/Transplant Oncologist Web Portal
  Shared Care: Shared Care involves four specific strategies to allow patients to have a portion of their care locally after HCT, where clinic and laboratory visits are equally shared between the local oncologist and primary HCT team
- Usual Care: * Patients receive all follow-up care at DFCI only, which is currently the Standard Care.
  * Majority of routine visits in first 180 days will be at DFCI.
  Standard Care: The usual care provided by the transplant center at DFCI.
Period: Overall Study
Arm/Group | Shared Care | Usual Care
Started | 166 | 160
Completed | 152 | 150
Not Completed | 14 | 10
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Transplant delayed or withdrawn | 12 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Shared Care | Usual Care | Total
Number analyzed (Participants) | 152 | 150 | 302
Age, Continuous [Median (Full Range); unit: years] | 63 [20 to 79] | 62 [20 to 77] | 63 [20 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 64 | 117
  Male | 99 | 86 | 185
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 141 | 136 | 277
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 8 | 12
Region of Enrollment [Number; unit: participants]
  United States | 152 | 150 | 302
Human leukocyte antigen (HLA) type [Count of Participants; unit: Participants]
  Matched Unrelated | 87 | 94 | 181
  Matched Related | 28 | 19 | 47
  Mismatched | 19 | 18 | 37
  Unknown/Other | 18 | 19 | 37

OUTCOME MEASURES:

1. Primary Outcome: Functional Assessment of Cancer Therapy - Bone Marrow Transplantation (FACT-BMT) at Day 180
Description: Functional Assessment of Cancer Therapy - Bone Marrow Transplantation TOTAL score. The TOTAL score is a summed combination of the Physical Well-Being (PWB), Social/Family Well-Being (SWB), Emotional Well-Being (EWB), Functional Well-Being (FWB) and Bone Marrow Transplant Subscales (BMTS). Higher scores (range: 0 - 148) represent better transplant-related quality of life. It was selected by a consensus of patient stakeholders as a patient-reported outcome (PRO) for the trial.
Time Frame: 180 days
Population: Participants with complete FACT-BMT responses sufficient to calculate the total FACT-BMT score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Shared Care | Usual Care
Number analyzed (Participants) | 86 | 86
score on a scale | 110.68 (18.34) | 106.89 (20.42)

2. Primary Outcome: European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire for Cancer (EORTC QLQ-C30) at Day 180
Description: European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire for Cancer GLOBAL health status subscale. Higher values (range: 0 to 100) represent higher quality of life. This was selected by a consensus of patient stakeholders.
Time Frame: 180 days
Population: Participants with complete EORTC QLQ-C30 response sufficient to calculate global score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Shared Care | Usual Care
Number analyzed (Participants) | 70 | 73
score on a scale | 68.93 (20.6) | 67.01 (20.76)

3. Primary Outcome: 100-day Non-relapse Mortality (NRM) for Patients in Shared Care Versus Usual Care
Description: Non-relapse mortality is a common measure to assess early outcomes for stem cell transplant, given that there can be a high level of early mortality from the transplant itself even in the absence of relapse. It is defined as a death occurring while in continuous remission. NRM is reported as a binary outcome.
Time Frame: 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | Shared Care | Usual Care
Number analyzed (Participants) | 152 | 150
Participants | 4 | 4

ADVERSE EVENTS:
Time Frame: Acute graft-versus-host disease (aGVHD), all-cause mortality and non-relapse mortality (NRM) was collected for the first 100 days of participation (until Day 100).
Description: Adverse event collection was limited to collection of aGVHD and NRM and graded on clinical scales. No other adverse events were collected.
Arm/Group | Shared Care | Usual Care
All-Cause Mortality (participants affected / at risk) | 9/152 | 7/150
Serious Adverse Events (participants affected / at risk) | 0/152 | 0/150
Other Adverse Events (participants affected / at risk) | 47/152 | 45/150
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Shared Care (N=152) | Usual Care (N=150)
Grade II-IV aGVHD D100 (Blood and lymphatic system disorders) | 26 (26) | 22 (22)
Grade I aGVHD D100 (Blood and lymphatic system disorders) | 21 (21) | 23 (23)

LIMITATIONS AND CAVEATS:
The Shared Care randomized clinical trial was limited by its status as a care delivery strategy wherein ability to share care with a local oncologist is heavily dependent on prevailing patient and participating center circumstances. Moreover, the study was not powered to detect QOL difference at earlier timepoints than Day 180.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-16): https://cdn.clinicaltrials.gov/large-docs/26/NCT03244826/Prot_SAP_000.pdf